CLINICAL TRIAL: NCT01173341
Title: Cardiotoxicity of Cancer Therapy: Mechanisms and Predictors
Brief Title: Cardiotoxicity of Cancer Therapy (CCT)
Status: Enrolling by invitation | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 09110
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Chemotherapy-induced cardiotoxicity; Anthracycline; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subgroup 2: Subgroup2 represents will undergo trastuzumab therapy only
  Interventions: Diagnostic Test: Echocardiography; Other: Blood Collection; Other: Symptoms Questionnaire
- Subgroup 1: Subgroup 1 are anthracycline only treated patients.
  Interventions: Diagnostic Test: Echocardiography; Other: Blood Collection; Other: Symptoms Questionnaire
- Subgroup 3: Subgroup 3 are patients that will undergo trastuzumab therapy with anthracyclines.
  Interventions: Diagnostic Test: Echocardiography; Other: Blood Collection; Other: Symptoms Questionnaire

INTERVENTIONS:
Diagnostic Test: Echocardiography — Prior to chemotherapy, prior to and after anthracyclines, every 6 weeks during trastuzumab, and yearly for up to 10 years.
Other: Blood Collection — Drawn at first chemo treatment and periodically during treatment (exact schedule varies with clinically ordered treatment plan), then annually for up to 10 years. Blood is banked for future biomarker testing.
Other: Symptoms Questionnaire — Survey collected at first chemotherapy, periodically during therapy (exact schedule determined by clinically ordered treatment regimen), and annually for up to 10 years.

SUMMARY:
The objective of this study is to define the clinical significance of mechanistic biomarkers (including Neuregulin-1Beta) and novel echocardiographic measures of cardiac function in predicting the incident risk of cancer therapy cardiotoxicity.

DETAILED DESCRIPTION:
The overall study objectives are:

1. To determine the longitudinal relationships between circulating markers, such as Neuregulin (NRG)-1Beta levels and incident risk of adverse cardiovascular outcomes in patients exposed to anthracycline, trastuzumab, or a combination of the two agents. We hypothesize that a sustained increase in NRG-1Beta, indicative of enhanced cardiac stress with exposure to chemotherapeutic agents, is predictive of an increased risk of cardiac dysfunction and heart failure.
2. To study the single nucleotide polymorphism (SNP)/haplotype variation in pathways of interest, such as the Neuregulin/Epidermal Growth Factor (ErbB) signaling pathway, on incident risk of adverse cardiovascular outcomes. We hypothesize that there will be SNP/haplotypes variations that are associated with incident cardiovascular outcomes.
3. To determine the longitudinal relationships between novel echocardiographic measures, such as strain and strain rate and incident cardiac dysfunction in patients exposed to anthracycline, trastuzumab, or a combination of the two agents. We hypothesize that early declines in strain and strain rate are predictive of an increased risk of future cardiac dysfunction and heart failure.
4. To explore the changes in biomarkers such as NRG-1Beta levels and the relationships with novel echocardiographic measures of cardiac function.
5. To create a biobank as a future resource for additional questions in novel biomarkers and genetics.
6. To determine the long-term effects of cancer therapy cardiotoxicity by following patients yearly for 5 years after their exposure to cancer therapy, with the option to extend up to an additional 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HER-2 positive breast cancer designated to receive trastuzumab chemotherapy with or without prior exposure to anthracycline-based chemotherapy
* Non-HER-2 positive breast cancer designated to receive treatment with an anthracycline-containing regimen

Exclusion Criteria:

* Other contraindications to trastuzumab or anthracycline chemotherapy.
* Vulnerable populations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with breast cancer will enter the cohort prior to chemotherapy initiation and be evaluated at baseline and at regular intervals during the first approximately 15 months after chemotherapy is initiated. Patients will have study visits at 2 years, 3 years, 5, years, 7 years, 9 years, 11 years, 13 years, and 15 years following initiation of cancer therapy.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2010-07 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Cardiac dysfunction or signs or symptoms of heart failure | 15 years
  Cardiac dysfunction. as defined according to the Cardiac Review and Evaluation Committee (CREC) criteria as a decline in LVEF of 10% to less than 55% without signs or symptoms

SECONDARY OUTCOMES:
Change in quantitated Left Ventricular Ejection Fraction (LVEF) | 15 years
  Change in LVEF over the course of chemotherapy; incident diastolic dysfunction by echocardiography; the combined endpoint of any incident adverse cardiovascular outcome (arrhythmia, heart failure, systolic dysfunction, or diastolic dysfunction by echo)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Demissei BG, Hubbard RA, Zhang L, Smith AM, Sheline K, McDonald C, Narayan V, Domchek SM, DeMichele A, Shah P, Clark AS, Fox K, Matro J, Bradbury AR, Knollman H, Getz KD, Armenian SH, Januzzi JL, Tang WHW, Liu P, Ky B. Changes in Cardiovascular Biomarkers With Breast Cancer Therapy and Associations With Cardiac Dysfunction. J Am Heart Assoc. 2020 Jan 21;9(2):e014708. doi: 10.1161/JAHA.119.014708. Epub 2020 Jan 21. PMID 31959034
- [Derived] Upshaw JN, Finkelman B, Hubbard RA, Smith AM, Narayan HK, Arndt L, Domchek S, DeMichele A, Fox K, Shah P, Clark A, Bradbury A, Matro J, Adusumalli S, Carver JR, Ky B. Comprehensive Assessment of Changes in Left Ventricular Diastolic Function With Contemporary Breast Cancer Therapy. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 2):198-210. doi: 10.1016/j.jcmg.2019.07.018. Epub 2019 Sep 18. PMID 31542526
- [Derived] Garcia-Pavia P, Kim Y, Restrepo-Cordoba MA, Lunde IG, Wakimoto H, Smith AM, Toepfer CN, Getz K, Gorham J, Patel P, Ito K, Willcox JA, Arany Z, Li J, Owens AT, Govind R, Nunez B, Mazaika E, Bayes-Genis A, Walsh R, Finkelman B, Lupon J, Whiffin N, Serrano I, Midwinter W, Wilk A, Bardaji A, Ingold N, Buchan R, Tayal U, Pascual-Figal DA, de Marvao A, Ahmad M, Garcia-Pinilla JM, Pantazis A, Dominguez F, John Baksi A, O'Regan DP, Rosen SD, Prasad SK, Lara-Pezzi E, Provencio M, Lyon AR, Alonso-Pulpon L, Cook SA, DePalma SR, Barton PJR, Aplenc R, Seidman JG, Ky B, Ware JS, Seidman CE. Genetic Variants Associated With Cancer Therapy-Induced Cardiomyopathy. Circulation. 2019 Jul 2;140(1):31-41. doi: 10.1161/CIRCULATIONAHA.118.037934. Epub 2019 Apr 16. PMID 30987448